CLINICAL TRIAL: NCT03006133
Title: Prevalence of Bruxism in a Group of Preschool Egyptian Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Wafik Ismael Mohamed, Demonstrator, Cairo University
Other Study IDs: CEBC-CU-2016-12-171
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The protocol is to show the prevalence of bruxism among a group of Egyptian children

DETAILED DESCRIPTION:
Many studies are done on children to show the prevalence of bruxism among different ages , reports of prevalence range from 8-31% in the general population, the prevalence of bruxism in Egyptian children is unknown. Several symptoms are commonly associated with bruxism, including hypersensitive teeth, aching jaw muscles, headaches, tooth wear, damage to dental restorations (e.g. crowns and fillings) and damage to teeth. However it may cause minimal symptoms, and therefore people may not be aware of the condition,so this study is important to determine the prevalence of bruxism of preschool Egyptian children

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative children from 3-6 years
2. Children without any Medical problems
3. Children of families who accept to participate in the study

Exclusion Criteria:

1- Children with caries in posterior teeth

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preschool Egyptian children
Sampling Method: Probability Sample
Enrollment: 362 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Bruxism | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Manal Ahmed, Cairo Governorate, Manial, Egypt